CLINICAL TRIAL: NCT02905825
Title: Clinical Confirmation Study to Confirm Safety and Presence of H. Pylori With 13C-Urea Breath Test Using the BreathID® Hp and BreathID® Hp Lab Systems in the Pediatric Population
Brief Title: Urea Breath Test (UBT) With Breath Hp System /BreathID Hp Lab System Pediatrics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PED-HP-0616B
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2018-06

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Occult Blood

STUDY DESIGN:
Intervention Model Description: A 13C labeled substrate is used as part of a combination product; a diagnostic breath test.
Masking Description: The investigator and treating physician will remain blinded to the breath test results until the end of the study. There is only one arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Indication for Helicobacter pylori testing (Experimental): Walk in basis: any pediatric subjects with indication for Helicobacter pylori testing will be enrolled if they meet study eligibility criteria and will perform stool test and urea breath test within a week of each other.
  Interventions: Device: BreathID® Hp System; Drug: BreathID® Hp Lab System; Diagnostic Test: Stool Test

INTERVENTIONS:
Device: BreathID® Hp System — Breath will be analyzed for change in carbon 13 content in breath after ingestion of carbon 13 enriched urea
Drug: BreathID® Hp Lab System — Breath will be analyzed for change in carbon 13 content in breath after ingestion of carbon 13 enriched urea
Diagnostic Test: Stool Test — Each subject was asked to perform a stool test in parallel to the breath test.
  Other Names: Stool Antigen Test

SUMMARY:
Clinical Study to Confirm Safety and Accuracy in Detection of H. pylori with 13C-Urea Breath Test using the BreathID® Hp and BreathID® Hp Lab Systems in the Pediatric Population

DETAILED DESCRIPTION:
Pediatric subjects with indication for H.pylori testing, will be tested with both stool antigen as a reference standard and a urea breath test using the BreathID® Hp and BreathID® Hp Lab Systems. The BreathID® Hp system continuously measures breath via a nasal cannula and the BreathID® Hp Lab System measures breath collection bags before and after ingestion of a solution with enriched carbon 13 urea and citric acid. The stool sample will be provided within a week of the breath tests and will be analyzed by a central laboratory. Safety and overall efficacy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Be older than 3 and younger than 18 years of age
* Present with a clinical indication compatible with H. pylori based on the judgement of the treating physician (such as abdominal pain, nausea, diarrhea, reflux, peptic ulcer, dyspepsia, etc., or following treatment for H.pylori)
* Subject/Legal guardian (and subject whenever relevant) is willing to sign the Informed Consent/Assent Form
* Naïve to H. pylori treatment in the past 6 weeks

Exclusion Criteria:

* Participation in other interventional trials
* PPI or H2 blockers within two (2) weeks prior to breath test/stool antigen test
* Pregnant or breastfeeding female
* Allergy to test substrates
* Antibiotics (not related to H. pylori eradication) and/or Bismuth preparations within four (4) weeks prior to breath test
* Exposure to any type of anesthesia, analgesics or sedation 24 hours prior to the breath test.
* Exposure to any 13C-enriched substance 24 hours prior to the breath test.
* Children 12 years and older - to be excluded after a written notification from the sponsor is received at the site that the limit of 1/3 of the sample size was achieved for this group
* Subjects outside US - to be excluded after a written notification from the sponsor is received at the site that the limit of 1/3 of the sample size was achieved for this group

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Willis-Knighton Pediatric GI Specialist/Willis-Knighton Physician Network, Shreveport, Louisiana
  - Gastrointestinal Associates, Flowood, Mississippi
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Health - Children's Medical Center Dallas (UT Southwestern), Dallas, Texas
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
- Assaf Harofe Medical Center, Tzrifin, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject (or parent) signed the consent, but before washout period was completed, decided to withdraw from trial. Therefore, from the 54 consented, only 53 started the study procedure.
Period: Overall Study
Arm/Group | Indication for Helicobacter Pylori Testing
Started | 53
Completed | 41
Not Completed | 12
Not completed — Protocol Violation | 11
Not completed — Device Malfunction | 1

BASELINE CHARACTERISTICS:
Arm/Group | Indication for Helicobacter Pylori Testing
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 53
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 37
  Israel | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reported Adverse Events
Description: Number of participants with reported adverse events after performing urea breath test
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Indication for Helicobacter Pylori Testing
Number analyzed (Participants) | 53
Participants | 1

2. Secondary Outcome: Percentage of Agreement
Description: Percentage of agreement between stool test reference standard and continuous urea breath test in assessing presence or absence of Helicobacter pylori infection
Time Frame: 1 week
Population: Although 42 subjects completed the protocol, there was a device malfunction in this arm, therefore only 41 performed the continuous test.
Measure: Number (95% Confidence Interval); unit: percentage of pos. or neg. agreeement
Arm/Group | Indication for Helicobacter Pylori Testing
Number analyzed (Participants) | 41
percentage of pos. or neg. agreeement | 97.56 [87.14 to 99.94]

3. Secondary Outcome: Percentage of Agreement
Description: Percentage of agreement between stool test reference standard and breath bags from urea breath test in assessing presence or absence of Helicobacter pylori infection
Time Frame: 1 week
Measure: Number (95% Confidence Interval); unit: percentage of pos. or neg. agreeement
Arm/Group | Indication for Helicobacter Pylori Testing
Number analyzed (Participants) | 42
percentage of pos. or neg. agreeement | 97.62 [87.43 to 99.94]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Indication for Helicobacter Pylori Testing
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 1/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indication for Helicobacter Pylori Testing (N=53)
Vomiting (Gastrointestinal disorders) | 1 (1) — Vomiting possibly induced by drinking of test substrate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the Proprietary Data in scientific journals and other scientific and professional publications and oral dissertations and the like, provided that a draft of the intended publication or dissertation shall be submitted to the Company at least sixty (60) days before the date of intended publication or dissertation so as to enable the Company to make comments to the Center regarding the contents of such intended publication or dissertation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT02905825/Prot_SAP_000.pdf